CLINICAL TRIAL: NCT01656304
Title: Phase II Trial of Bevacizumab in PSA Relapse Androgen Independent Prostate Cancer (AVF3952sn)
Brief Title: Bevacizumab in Treating Patients With Relapsed Prostate Cancer That Did Not Respond to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Ulka Vaishampayan, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-064; NCI-2011-00661 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCT00478413 (obsolete NCT alias)
Record Dates: First submitted 2012-07-30; First posted 2012-08-02 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (monoclonal antibody, antiangiogenesis) (Experimental): Patients receive bevacizumab IV over 30-90 minutes once every 14 days. Courses repeat every 14 days in the absence of disease progression and unacceptable toxicity.
  Interventions: Biological: bevacizumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot phase II trial studies how well giving bevacizumab works in treating patients with relapsed prostate cancer that did not respond to hormone therapy. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or tumor-killing substances to them. Bevacizumab may also stop the growth of prostate cancer by blocking blood flow to the tumor

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The rate of prostate-specific antigen (PSA) response with avastin (bevacizumab) therapy in androgen independent non-metastatic prostate cancer.

II. Toxicities associated with avastin therapy. III. Time to PSA progression.

SECONDARY OBJECTIVES:

I. Overall survival of androgen independent non-metastatic prostate cancer patients treated with avastin.

II. The change in PSA velocity with avastin therapy in androgen-independent non-metastatic prostate cancer.

III. Time to distant metastatic disease. IV. Circulating tumor cell count. V. Changes in levels of N terminal collagen peptide and bone-specific alkaline phosphatase with avastin therapy.

VI. Correlation of crosslinked N-telopeptide of type I collagen (NTX) and serum B-Cell-Specific Activator Protein (BSAP) levels with time to PSA progression.

OUTLINE:

Patients receive bevacizumab intravenously (IV) over 30-90 minutes once every 14 days. Courses repeat every 14 days in the absence of disease progression and unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* A histologic diagnosis of prostate adenocarcinoma.
* No evidence of bone/visceral metastases as visualized on standard imaging such as bone scan, chest X-ray, CT scan or MRI of abdomen and pelvis.
* PSA-only progression despite androgen deprivation therapy. PSA progression is defined as 3 rising levels, with a minimum interval of 2 weeks between each determination. The last determination must have a minimum value of

  1ng/ml and be determined within two weeks prior to registration. If the second or third confirmatory value is less than the previous value, the patient will still be eligible if a repeat value (No. 4) is found to be greater than all the prior values.
* If patient has been on antiandrogen in the past 28 days, then PSA progression after withdrawal period (28 days for flutamide and 42 days for bicalutamide or nilutamide) is required.
* ECOG performance status of 0-1.
* No prior avastin therapy.
* No investigational or commercial agents or therapies (except LHRH agonists) may be administered concurrently with the intent to treat the patient's malignancy. Patients on LHRH agonists must continue the use of LHRH agonist therapy. Bisphosphonates can be administered per treating physician discretion.
* At least 4 weeks must have elapsed since prior systemic therapy, except for LHRH analogue therapy and steroids. If steroids are being used for therapy of prostate cancer, these should be discontinued prior to starting avastin therapy.
* Age ≥ 18 years.
* Life expectancy of at least 6 months.
* Ability to understand and the willingness to sign a written informed consent that is approved by the Institutional Human Investigation Committee.
* Use of effective means of contraception in subjects.

Exclusion Criteria:

Inability to comply with study and/or follow-up procedures.

* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications).
* Any prior history of hypertensive crisis or hypertensive encephalopathy.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix E).
* History of myocardial infarction or unstable angina within last 12 months prior to study enrollment.
* History of stroke or transient ischemic attack within 6 months prior to study enrollment.
* Known CNS disease.
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection).
* Symptomatic peripheral vascular disease.
* Evidence of bleeding diathesis or coagulopathy.
* Patients on anticoagulants are allowed if patient has been on therapy for at least 4 weeks and patient has no acute thromboembolic activity.
* Major surgical procedure, open biopsy, or significant traumatic injury within. 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study.
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment.
* Serious, non-healing wound, ulcer, or bone fracture.
* Proteinuria at screening as demonstrated by:

  1. Urine protein:creatinine (UPC) ratio ≥ 1.0 at screening
* Known hypersensitivity to any component of avastin.
* Refusal to use effective means of contraception.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to avastin.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with immune deficiency such as HIV-positive patients or those receiving combination anti-retroviral therapy are excluded from the study because of lack of safety data for avastin in these patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-05; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulka Vaishampayan, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Monoclonal Antibody, Antiangiogenesis)
Started | 16
Completed | 15
Not Completed | 1
Not completed — Ineligible, uncontrolled hypertension | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Monoclonal Antibody, Antiangiogenesis)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.53 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: PSA Response Rate With Bevacizumab Therapy in Androgen Independent Non-metastatic Prostate Cancer
Description: A PSA response will be considered a PSA decline of at least 50% must be confirmed by a second PSA value four or more weeks later. The reference PSA for these declines should be a PSA measured within 2 weeks prior to the initiation of therapy. Response rates will be summarized by point estimates and Wilson type 80% confidence intervals.
Time Frame: An average every 6 weeks for up to 3 months
Measure: Number; unit: participants
Arm/Group | Treatment (Monoclonal Antibody, Antiangiogenesis)
Number analyzed (Participants) | 15
participants | 5
Statistical Analysis 1: Comparison: Treatment (Monoclonal Antibody, Antiangiogenesis); Test type: Superiority or Other; Rate = .333, 80% CI 2-sided [.20 to .50], Standard Error of Mean .1217

2. Primary Outcome: Toxicities Associated With Bevacizumab Therapy
Description: Toxicity rates will be summarized by point estimates and Wilson type 90% confidence intervals. Toxicities will be graded per the National Cancer Institute (NCI) Common Toxicity Criteria (CTC), and PSA response will be determined as per PSA Working Group response criteria. Censored time to PSA progression will be estimated with standard Kaplan-Meier methodology.
Time Frame: An average of every 2 weeks while on therapy
Measure: Number; unit: participants
Arm/Group | Treatment (Monoclonal Antibody, Antiangiogenesis)
Number analyzed (Participants) | 15
participants | 14

3. Primary Outcome: Time to PSA Progression (TTPP)
Description: TTPP will be measured from protocol registration to appearance of PSA progression as defined by the criteria of the PSA Working Group response criteria. The end point for progression will be calculated at the time a 25% increase in PSA has been achieved. PSA velocity will also be calculated as change in PSA doubling time pre and post therapy and the rate of PSA rise pre- and post-therapy.
Time Frame: An average every 6 weeks for up to 3 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Monoclonal Antibody, Antiangiogenesis)
Number analyzed (Participants) | 15
months | 2.8 [2.4 to 5.4]

4. Secondary Outcome: Overall Survival of Androgen Independent Non-metastatic Prostate Cancer Patients Treated With Bevacizumab
Description: Overall survival of androgen independent non-metastatic prostate cancer patients treated with bevacizumab. The number of patients still alive at the end of the study (median K-M estimate cannot be obtained due to the 86.7% censoring rate).
Time Frame: Every 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Monoclonal Antibody, Antiangiogenesis)
Number analyzed (Participants) | 15
Participants | 13

5. Secondary Outcome: The Change in PSA Velocity With Bevacizumab Therapy in Androgen Independent Non-metastatic Prostate Cancer
Description: PSA velocity with bevacizumab therapy in androgen independent non-metastatic prostate cancer pre-therapy, as well as, PSA velocity with bevacizumab therapy while on therapy.
Time Frame: Baseline, every 6 weeks while on therapy, and then every 3 months thereafter
Measure: Median (Full Range); unit: ng/ml/month
Arm/Group | Treatment (Monoclonal Antibody, Antiangiogenesis)
Number analyzed (Participants) | 15
ng/ml/month
  Pre-therapy | 2.64 [0.29 to 37.07]
  On therapy | 1.87 [0.22 to 16.15]

6. Secondary Outcome: Time to Distant Metastatic Disease
Description: Time to distant metastatic disease using the Kaplan-Meier method
Time Frame: Every 3 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Monoclonal Antibody, Antiangiogenesis)
Number analyzed (Participants) | 15
months | 7.9 [3.2 to 17.6]

ADVERSE EVENTS:
Arm/Group | Treatment (Monoclonal Antibody, Antiangiogenesis)
Serious Adverse Events (participants affected / at risk) | 4/16
Other Adverse Events (participants affected / at risk) | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Monoclonal Antibody, Antiangiogenesis) (N=16)
Hypertension (Vascular disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Monoclonal Antibody, Antiangiogenesis) (N=16)
ALT increase (Investigations) | 1 (1)
AST Increase (Investigations) | 2 (2)
GERD (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Edema (General disorders) | 1 (1)
Elevated Creatinine (Investigations) | 2 (2)
Fatigue (General disorders) | 7 (7)
Generalized Pain (General disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Hemorrhage GI (Gastrointestinal disorders) | 1 (1)
Hemorrhage GU (Gastrointestinal disorders) | 1 (1)
Hemorrhage GU-prostate/urethra (Gastrointestinal disorders) | 1 (1)
Hemorrhage nose (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemorrhage oral cavity (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Leukopenia (Investigations) | 1 (1)
Lower Extremity swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 6 (6)
Thrombocytopenia (Investigations) | 1 (1)
Urine color change (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
weight loss (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
There was a small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No